CLINICAL TRIAL: NCT01974986
Title: Rehydration Following Exercise-Induced Dehydration: Beverage Formula Effects in Team Sport Athletes
Brief Title: Rehydration Following Exercise-Induced Dehydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Principal Investigator, Craig A. Horswill, Clinical Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AN-US-1307
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Dehydration Related to Exercise
Keywords: dehydration; exercise; rehydration; sodium; water; carbohydrate
MeSH Terms: conditions — Dehydration; Motor Activity | interventions — Water; Flavoring Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Water with flavoring and non-nutritive sweetener.
  Interventions: Other: Water with flavoring and non-nutritive sweetener.
- High-Na low-CHO beverage (Experimental): Beverage containing sodium concentration of 40 to 50 mEq/L and carbohydrate concentration between 310 and 350 mmol/L.
  Interventions: Other: High-Na low-CHO beverage
- Low-Na high-CHO beverage (Experimental): Beverage containing sodium concentration of 15 to 25 mEq/L and carbohydrate concentration between 120 and 160 mmol/L.
  Interventions: Other: Low-Na high-CHO beverage

INTERVENTIONS:
Other: Water with flavoring and non-nutritive sweetener. — A volume of fluid (water) was given after exercise to return each subject's body mass (to euhydration).
  Arms: Placebo
Other: High-Na low-CHO beverage — A volume of fluid (high-Na, low-CHO) was given after exercise to return each subject's body mass (to euhydration).
  Arms: High-Na low-CHO beverage
Other: Low-Na high-CHO beverage — A volume of fluid (low-Na, high-CHO) was given after exercise to return each subject's body mass (to euhydration).
  Arms: Low-Na high-CHO beverage

SUMMARY:
Athletes participating in multiple training sessions a day can be at increased risk of suboptimal hydration and heat illness during their second training session, especially when the environment is hot and humid. With the exception of the absolute volume of water delivered by a rehydration beverage, characteristics of the beverage consumed play a role in the recovery and completeness of rehydration. The amount of sodium in the beverage has been shown to be a primary factor in rehydration. Recently, an effect of the carbohydrate concentration of the beverage was been reported, with its effects mediated by the renal system in response to elevated serum insulin. The purpose of this study is to compare sodium and carbohydrate effects on rehydration and recovery.

DETAILED DESCRIPTION:
The effectiveness of beverage composition will be evaluated by modifying the sodium content and carbohydrate content of the beverage. Hypothesis: Completeness of rehydration will be greater in the beverage with higher sodium concentration. It is also hypothesized that electrolyte-carbohydrate beverages will promote rehydration that exceeds that of consuming placebo (water). Using a randomized balanced-treatment crossover design, physically trained males (18-35 yrs) will participate in intermittent exercise for 85 to 100 minutes in three experimental trials of variable intensity training in the heat (30 +/-3 C) followed by a rehydration-recovery period. Exercise will be done at varying intensities (intermittent intervals) ranging from 50% to nearly 100% of maximum oxygen uptake (max VO2) determined prior to the experimental trials. During the 85 to 100 min of exercise, no fluids will be given during the trial to elicit an acute reduction in body mass of approximately 2.5 to 3% (standardized for each subject). Following exercise, 100% of the volume of fluid lost will be replaced with one of the beverages. Beverages will be ingested in six aliquots over a 1-hr period given at the end of the trial. Retention of fluid will be calculated by measuring volume of urine lost at 30, 60, 135, and 210 min following ingestion of the rehydration beverage. The primary outcome variable is the percentage of fluid retained, i.e., the difference between volume ingested and cumulative urine produced in 3.5 h as a percentage of volume ingested. Body mass, urine specific gravity, total body water, and ratings of vigor and affect will be assessed prior to exercise, after exercise in a state of dehydration, and at 210 min post-exercise following rehydration. A one-way ANOVA will be used to test the hypothesis for rehydration, the primary outcome variable.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18-35 y, physically fit, and regularly undergoing exercise training particularly but not exclusively in team sports.

Exclusion Criteria:

* "Yes" on PAR-Q survey, symptoms or signs of exercise intolerance, VO2 max <50 mL/kg/min, smoker

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Rehydration | 8 hours
  Fluid retained to rehydrate the body as a percentage of volume of beverage ingested.

SECONDARY OUTCOMES:
Body weight | 8 hours
  Change in body mass from the start of data collection.

OTHER OUTCOMES:
Total body water | 8 hours
  Change in estimated total body water from the start of data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Horswill, PhD, Principal Investigator — UIC
Locations (1):
- University of Illinois, Chicago, Illinois, United States